CLINICAL TRIAL: NCT04051307
Title: Dual Vaccine Trial in Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Prof, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPN19H2
Record Dates: First submitted 2019-07-11; First posted 2019-08-09 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): Vaccination with:
  PD-L1 peptide:
  PD-L1 Long(19-27) Peptide sequence: FMTYWHLLNAFTVTVPKDL Dose: 100 µg PD-L1 long1 dissolved in DMSO/water - Total volume: 0,5 ml.
  Arginase1 peptide:
  ArgLong2(169-206) Peptide sequence ISAKDIVYIGLRDVDPGEHYILKTLGIKYFSMTEVDRL Dose: 200 µg ARGLong2 dissolved in DMSO/water - Total volume: 0,5 ml.
  Both vaccines are given at a treatment. Adjuvant Montanide ISA 51 0,5ml is mixed with the peptides before treatment To be administered every second week - a total of twelve times, with a possibility of additional six treatments.
  Interventions: Drug: PD-L1 peptide: PD-L1 Long(19-27) Peptide sequence: FMTYWHLLNAFTVTVPKDL; Drug: Arginase1 peptide: ArgLong2(169-206) Peptide sequence ISAKDIVYIGLRDVDPGEHYILKTLGIKYFSMTEVDRL

INTERVENTIONS:
Drug: PD-L1 peptide: PD-L1 Long(19-27) Peptide sequence: FMTYWHLLNAFTVTVPKDL — Peptide vaccination
  Other Names: PD-L1Long
Drug: Arginase1 peptide: ArgLong2(169-206) Peptide sequence ISAKDIVYIGLRDVDPGEHYILKTLGIKYFSMTEVDRL — Peptide vaccination
  Other Names: ARGLong2

SUMMARY:
A phase I-II study in patients with mutated MPN by vaccinating with PD-L1 and Aginase1 peptides with Montanide ISA-51 as adjuvant, to monitor the immunological response to vaccination and subsequently safety, toxicity and clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of essential thrombocythemia or Polycythemia Vera, according to the WHO criteria123,124 2. Age ≥18 years 3. Performance status ≤ 2 (ECOG-scale) 4. Expected survival > 3 months 5. Sufficient bone marrow function 6. Creatinine < 2.5 upper normal limit, i.e. < 300 µmol/l 7. Sufficient liver function, i.e.

  1. ALAT < 2.5 upper normal limit, i.e. ALAT <112 U/l
  2. Bilirubin < 30 U/l 8. For women: Agreement to use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 120 days after the last treatment.

     9. For men: Agreement to use contraceptive measures and agreement to refrain from donating sperm.

     Exclusion criteria
     1. Other malignancies in the medical history excluding basal cell carcinoma. Patients cured for another malignant disease with no sign of relapse five years after ended treatment is allowed to enter the protocol.
     2. Significant medical condition per investigators judgement e.g. severe Asthma/COPD, poorly regulated heart condition, insulin dependent diabetes mellitus.
     3. Acute or chronic viral or bacterial infection e.g. HIV, hepatitis or tuberculosis
     4. Serious known allergies or earlier anaphylactic reactions.
     5. Known sensibility to Montanide ISA-51
     6. Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
     7. Pregnant and breastfeeding women.
     8. Fertile women not using secure contraception with a failure rate less than < 1%
     9. Patients taking immune suppressive medications incl. systemic corticosteroids and methotrexate at the time of enrollment
     10. Psychiatric disorders that per investigator judgment could influence compliance.
     11. Treatment with other experimental drugs
     12. Treatment with other anti-cancer drugs - except IFN-a, hydroxyurea or anagrelide.
     13. Treatment with ruxolitinib.
     14. Treatment with chemotherapy or immune therapy (excluding IFN-a, hydroxyurea or anagrelide) within the last 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Immune response | 1 year
  T-cell cytokine release towards target antigens

SECONDARY OUTCOMES:
Adverse events evaluated by CTCAE v. 5.0 | 1 year
  Adverse events are graded 1-5 according to the criteria
Clinical response | 10 year
  Vaccinations will induce clinical response in 2 patients, either partial response or better, according response criteria for PV and ET or clinical response as a reduction of mutated allelic burden - 10% from baseline at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob H Grauslund, MD, Principal Investigator — CENTER FOR CANCER IMMUNE THERAPY, CCIT-DK
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev, Capital Region
  - National Center for Cancer Immune Therapy (CCIT-DK), Herlev

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grauslund JH, Holmstrom MO, Martinenaite E, Lisle TL, Glockner HJ, El Fassi D, Klausen U, Mortensen REJ, Jorgensen N, Kjaer L, Skov V, Svane IM, Hasselbalch HC, Andersen MH. An arginase1- and PD-L1-derived peptide-based vaccine for myeloproliferative neoplasms: A first-in-man clinical trial. Front Immunol. 2023 Feb 23;14:1117466. doi: 10.3389/fimmu.2023.1117466. eCollection 2023. PMID 36911725